CLINICAL TRIAL: NCT01835132
Title: Gevokizumab Treatment for Active Scleritis By IL-1 Inhibition (GATSBY)
Brief Title: Gevokizumab for Active Scleritis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Collaborators: The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 130102; 13-EI-0102 (Other: NIH CNS IRB)
Record Dates: First submitted 2013-04-16; First posted 2013-04-18 (Estimated); Results first posted 2015-08-25 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2017-10

CONDITIONS: Scleritis
Keywords: Scleritis; IL-1
MeSH Terms: conditions — Scleritis

STUDY DESIGN:
Intervention Model Description: Subcutaneous injection of 60 mg gevokizumab
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gevokizumab (Experimental): Subcutaneous injection of 60 mg gevokizumab
  Interventions: Device: Gevokizumab

INTERVENTIONS:
Device: Gevokizumab — Subcutaneous injection of 60 mg gevokizumab

SUMMARY:
Background:

- Scleritis is the inflammation of the white outer coating of the eye, known as the sclera. In severe cases, it can cause blindness. It is commonly associated with autoimmune disorders such as rheumatoid arthritis. Mild scleritis can be treated with drugs such as ibuprofen. More severe scleritis may need oral steroids or immunosuppressive treatments; however, these treatments can cause side effects in the whole body. Gevokizumab is a newer anti-inflammatory drug that is under investigation to treat other inflammatory diseases. It may not have as severe side effects as some other drugs. However, it has not yet been used to treat scleritis. Researchers want to see if it can be given as a safe and effective treatment for scleritis.

Objectives:

- To see if gevokizumab is a safe and effective treatment for scleritis.

Eligibility:

- Individuals at least 18 years of age who have active scleritis.

Design:

* There is an initial phase and a two-part extension phase in this study. The extension phase is optional. The initial phase of the study requires seven visits to the National Eye Institute (NEI).
* Participants will be screened with a physical exam and eye exam, and medical history will be obtained. Blood and urine samples will be collected.
* Eligible participants will receive an injection of 60 mg of gevokizumab at the first study visit and at Weeks 4, 8, and 12. They will be given under the skin by the stomach, or in the upper arm or thigh.
* Participants will have additional visits after the first study visit at Weeks 2, 16, and 28. No injection will be given at these visits. Eye exams will be done, and blood and tear samples will be collected.
* If the scleritis improves by Week 16, participants may choose to continue the study in the extension phase. In the 1st extension, they will have a visit every 4 weeks until Week 36 and then two additional monitoring visits at Weeks 40 and 52 for a total of 13 study visits.
* Participants who are eligible at Week 52 may continue in the "as needed" (PRN) extension phase (2nd extension) and receive gevokizumab injections (60 mg) at Weeks 52, 54, 58 and 62.

DETAILED DESCRIPTION:
Objective: Scleritis is a chronic, painful and potentially blinding inflammatory disease characterized by edema of the episcleral and sclera tissues and is commonly associated with systemic autoimmune disorders. Gevokizumab is an interleukin-1β (IL-1β) inhibitor, thus possibly preventing the IL-1β that may be responsible for scleral breakdown in patients with anterior scleritis. The study objective is to evaluate the safety and potential efficacy of gevokizumab as a possible treatment of non-infectious, active, anterior scleritis.

Study Population: Ten participants with non-infectious, active, anterior scleritis with a scleral inflammatory grade of ≥ +1 in at least one eye were to be initially enrolled. However, only eight participants were enrolled. Participants may be on ≤ 20 mg/day of prednisone or the equivalent at the time of enrollment but all other immunosuppressive drugs will be stopped with the initiation of study drug.

Design: This is a Phase 1/2, open label, non-randomized, prospective, single-arm, pilot trial to evaluate the safety and potential efficacy of gevokizumab in non-infectious, active, anterior scleritis. The study consists of an initial phase followed by a two-part extension phase. For the initial phase, all participants will receive one subcutaneous injection of 60 mg gevokizumab at Baseline and Weeks 4, 8 and 12. At Week 16 of the initial phase, participants will be assessed for eligibility in the first extension phase of the study. Participants from the initial phase, who do not continue in the first extension phase of the study will discontinue the study drug and may receive salvage therapy using standard-of-care treatment at the investigator's discretion. Participants from the initial phase who do not continue in the first extension phase will return for a final safety visit at Week 28. Participants from the initial phase who are determined eligible for the first extension phase may continue in the first extension phase and receive one gevokizumab injection (60 mg) every four weeks until the Week 36 visit. Participants entering the first extension phase will have follow-up safety visits at Weeks 40 and 52. At Week 52 follow-up of the first extension phase, participants will be assessed for eligibility in the 2nd extension phase, which is a PRN extension phase of the study. Participants who are eligible may continue in the PRN extension phase (2nd extension) and receive gevokizumab injections (60 mg) at Weeks 52, 54, 58, and 62. Subjects that have already completed the week 52 visit will be eligible to return and be assessed for entry into this 2nd extension phase. If they have already completed the Week 52 exit visit from the protocol and are returning to enroll in the PRN extension phase (2nd extension), the visits will be labeled as Weeks 52 (PRN-week0), 54 (PRN-week2), 58 (PRN-week6), and 62 (PRN-week10). Participants in the PRN extension phase (2nd extension) will have a final safety visit at least 16 weeks following their last injection in the PRN extension phase (2nd extension).

Outcome Measures: The primary outcome is the number of participants with at least a 2-step reduction or reduction to grade 0 in scleral inflammation in the study eye (or eyes, if both eyes meet study eye criteria), according to a standardized photographic scleritis grading system developed at NEI, on or before the Week 16 visit as compared to Baseline. Secondary outcomes include changes in visual acuity, changes in intraocular pressure and changes in scleral grading. Safety outcomes include the number and severity of systemic and ocular toxicities and adverse events (AEs), and the proportion of participants with loss of ≥ 15 ETDRS letters at any follow-up visit.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Participant must be 18 years of age or older.
2. Participant must have a diagnosis of non-infectious anterior scleritis requiring treatment.
3. Participant must agree not to undergo elective major surgery for the first 16 weeks of the study.
4. Participant must not have received any the following:

   * Another systemic biologic immunosuppressive agent within the last three months prior to enrollment (e.g., infliximab, daclizumab, etanercept, adalimumab, anakinra);
   * Rituximab or alkylating agent (e.g., cyclophosphamide) within the last 12 months prior to enrollment.
5. Participants on systemic anti-inflammatory therapy (including corticosteroids) must not have had a dose escalation in any of their immunosuppressive treatments within the last four weeks prior to enrollment.
6. Participant must stop all immunosuppressives upon enrollment in the study, with the exception of ≤ 20 mg/day of prednisone or equivalent.
7. Participant must have chest X-ray results (frontal and lateral) within the last 12 weeks prior to enrollment with no evidence of active pulmonary infection, active tuberculosis (TB) or malignancy.
8. Participant must be cleared by internal medicine for enrollment.
9. Female participants of childbearing potential must not be pregnant or breast-feeding, must have a negative pregnancy test at screening and must be willing to undergo pregnancy tests throughout the study.
10. Both female participants of childbearing potential and male participants able to father a child must have (or have a partner who has) had a hysterectomy or vasectomy, be completely abstinent from intercourse or must agree to practice two acceptable methods of contraception throughout the course of the study and for four months after the last investigational product injection. Acceptable methods of contraception include:

    * hormonal contraception (i.e., birth control pills, injected hormones, dermal patch or vaginal ring),
    * intrauterine device,
    * barrier methods (diaphragm, condom) with spermicide, or
    * surgical sterilization (tubal ligation).
11. Participant must be able to undergo slit lamp biomicroscopy on both eyes.
12. Participant must understand and sign the protocol's informed consent document.

EXCLUSION CRITERIA:

1. Participant has a significant active infection that requires treatment or has a history of recurrent systemic infections.
2. Participant has a history of TB and s/he has not received a full course of TB treatment, OR participant has a history of latent TB infection [or a positive Interferon-Gamma Release Assay (IGRA)] and has not received prophylactic treatment with isoniazid [also known as isonicotinylhydrazine (INH)] or rifampicin within the last six months prior to enrollment.
3. Participant is seropositive for human immunodeficiency virus (HIV) or Hepatitis C.
4. Participant has Hepatitis B. Positivity for Hepatitis B without evidence of active disease (per investigator judgment) is not exclusionary.
5. Participant has a history of cancer (other than a non-melanoma skin cancer or carcinoma in situ of the cervix) diagnosed within the last five years.
6. Participant has a history of severe allergic or anaphylactic reaction to monoclonal antibodies.
7. Participant has a history of previous treatment with gevokizumab.
8. Participant received live (attenuated) vaccine within the last three months prior to enrollment. Live seasonal flu and H1N1 vaccines are permitted ≥ two weeks prior to enrollment. Recombinant or killed vaccines are permitted at any time.
9. Participant has received an investigational drug or device within the last three months.
10. Participant has active joint or systemic inflammation requiring immediate addition or increase in systemic anti-inflammatory medications.
11. Participant has a condition (e.g., psychiatric illness, severe alcoholism or drug abuse) or situation that may put the participant at significant risk, may confound the study results or may interfere significantly with his/her participation or cooperation in the study.

STUDY EYE ELIGIBILITY CRITERIA:

The participant must have at least one eye meeting all inclusion criteria and none of the exclusion criteria listed below.

STUDY EYE INCLUSION CRITERIA:

1. Participant must have scleritis with a grade of ≥ +1 in the study eye.
2. Participant must have visual acuity of 20/640 or better in the study eye.
3. Participant must agree not to undergo elective ocular surgery (e.g., cataract extraction) in the study eye for the first 16 weeks of the study.

STUDY EYE EXCLUSION CRITERIA:

1. Participant has had any of the following in the study eye:

   * periocular, intravitreal steroid injection within the last six weeks prior to enrollment,
   * Ozurdex within the last six months prior to enrollment, or
   * Retisert within the last three years prior to enrollment.
2. Participant has had intraocular surgery in the study eye in the last four weeks prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-03; Primary Completion 2014-07 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hatice N Sen, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rothova A, Suttorp-van Schulten MS, Frits Treffers W, Kijlstra A. Causes and frequency of blindness in patients with intraocular inflammatory disease. Br J Ophthalmol. 1996 Apr;80(4):332-6. doi: 10.1136/bjo.80.4.332. PMID 8703885
- [Background] Jabs DA, Mudun A, Dunn JP, Marsh MJ. Episcleritis and scleritis: clinical features and treatment results. Am J Ophthalmol. 2000 Oct;130(4):469-76. doi: 10.1016/s0002-9394(00)00710-8. PMID 11024419
- [Background] Watson PG, Hayreh SS. Scleritis and episcleritis. Br J Ophthalmol. 1976 Mar;60(3):163-91. doi: 10.1136/bjo.60.3.163. PMID 1268179
- [Result] Knickelbein JE, Tucker WR, Bhatt N, Armbrust K, Valent D, Obiyor D, Nussenblatt RB, Sen HN. Gevokizumab in the Treatment of Autoimmune Non-necrotizing Anterior Scleritis: Results of a Phase I/II Clinical Trial. Am J Ophthalmol. 2016 Dec;172:104-110. doi: 10.1016/j.ajo.2016.09.017. Epub 2016 Sep 20. PMID 27663070
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-EI-0102.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Initial Phase: All participants have injections at Baseline, Wks 4, 8, and 12 with follow up visits at Wks 2, 16, and 28. 1st Extension Phase: If improved by Wk 16, visits every 4 wks until Wk 36 and then 2 visits at Wks 40 and 52. As-needed 2nd Extension Phase: At Week 52, if eligible, may continue with injections at Wks 52, 54, 58 and 62.
Period: Initial Phase
Arm/Group | Gevokizumab
Started | 8
Completed | 6
Not Completed | 2
Not completed — Insufficient Therapeutic Response | 2
Period: 1st Extension Phase
Arm/Group | Gevokizumab
Started | 6
Completed | 6 (Completed 52 Weeks)
Not Completed | 0
Period: 2nd Extension Phase - As Needed (PRN)
Arm/Group | Gevokizumab
Started | 3 (PRN extension - Participants starting this phase may not equal those who completed the 1st extension)
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gevokizumab
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 59.88 [34 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least a 2-step Reduction or Reduction to Grade 0 in Scleral Inflammation in the Study Eye (or Eyes), According to the National Eye Institute (NEI) Photographic Scleritis Grading System, on or Before the Week 16 Visit.
Description: Scleral inflammation was graded following 10% Phenylephrine application with an ordinal scale of 0 (no scleral inflammation with complete blanching of vessels), 0.5+ (minimal/trace inflammation with localized pink appearance of the sclera around minimally dilated deep episcleral vessels), 1+ (mild inflammation with diffuse pink appearance of the sclera around mildly dilated deep episcleral vessels), 2+ (moderate inflammation with purplish pink appearance of the sclera with tortuous and engorged deep episcleral vessels), 3+ (severe inflammation with diffuse significant redness of sclera, the details of superficial and deep episcleral vessels can't be observed), and 4+ (necrotizing inflammation with diffuse redness of the sclera with scleral thinning and uveal show).
Time Frame: Baseline and Week 16
Measure: Number; unit: participants
Arm/Group | Gevokizumab
Number analyzed (Participants) | 8
participants | 6

2. Secondary Outcome: Mean Change in Visual Acuity in the Study Eye (or Eyes) at Week 2 Compared to Baseline
Description: Visual acuity was measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol. Acuity is measured as letters read on an ETDRS eye chart and the letters read equate to Snellen measurements. For example, if a participant reads between 84 and 88 letters, the equivalent Snellen measurement is 20/20.
Time Frame: Baseline and Week 2
Population: Eight participants were active from Baseline to Week 28. Of the eight active participants, one participant had two study eyes, and this participant was active in the study to Week 28. A total of two participants did not continue past Week 28 due to insufficient therapeutic response. Six participants were active from Week 32 to Week 52.
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: eyes
Arm/Group | Gevokizumab
Number analyzed (Participants) | 8
Number analyzed (eyes) | 9
ETDRS letters | -1.00 (4.42)

3. Secondary Outcome: Mean Change in Visual Acuity in the Study Eye (or Eyes) at Week 4 Compared to Baseline
Description: as for outcome 2
Time Frame: Baseline and Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: eyes
Arm/Group | Gevokizumab
Number analyzed (Participants) | 8
Number analyzed (eyes) | 9
ETDRS letters | -1.78 (3.23)

4. Secondary Outcome: Mean Change in Visual Acuity in the Study Eye (or Eyes) at Week 8 Compared to Baseline
Description: as for outcome 2
Time Frame: Baseline and Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: eyes
Arm/Group | Gevokizumab
Number analyzed (Participants) | 8
Number analyzed (eyes) | 9
ETDRS letters | 0.78 (4.84)

5. Secondary Outcome: Mean Change in Visual Acuity in the Study Eye (or Eyes) at Week 12 Compared to Baseline
Description: as for outcome 2
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: eyes
Arm/Group | Gevokizumab
Number analyzed (Participants) | 8
Number analyzed (eyes) | 9
ETDRS letters | 0.11 (3.86)

6. Secondary Outcome: Mean Change in Visual Acuity in the Study Eye (or Eyes) at Week 16 Compared to Baseline
Description: as for outcome 2
Time Frame: Baseline and Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: eyes
Arm/Group | Gevokizumab
Number analyzed (Participants) | 8
Number analyzed (eyes) | 9
ETDRS letters | 1.00 (6.61)

7. Secondary Outcome: Mean Change in Visual Acuity in the Study Eye (or Eyes) at Week 20 Compared to Baseline
Description: as for outcome 2
Time Frame: Baseline and Week 20
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: eyes
Arm/Group | Gevokizumab
Number analyzed (Participants) | 8
Number analyzed (eyes) | 9
ETDRS letters | 1.33 (3.64)

8. Secondary Outcome: Mean Change in Visual Acuity in the Study Eye (or Eyes) at Week 24 Compared to Baseline
Description: as for outcome 2
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: eyes
Arm/Group | Gevokizumab
Number analyzed (Participants) | 8
Number analyzed (eyes) | 9
ETDRS letters | -0.67 (4.47)

9. Secondary Outcome: Mean Change in Visual Acuity in the Study Eye (or Eyes) at Week 28 Compared to Baseline
Description: as for outcome 2
Time Frame: Baseline and Week 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: eyes
Arm/Group | Gevokizumab
Number analyzed (Participants) | 8
Number analyzed (eyes) | 9
ETDRS letters | 1.00 (3.20)

10. Secondary Outcome: Mean Change in Visual Acuity in the Study Eye (or Eyes) at Week 32 Compared to Baseline
Description: as for outcome 2
Time Frame: Baseline and Week 32
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: eyes
Arm/Group | Gevokizumab
Number analyzed (Participants) | 6
Number analyzed (eyes) | 6
ETDRS letters | 3.00 (3.90)

11. Secondary Outcome: Mean Change in Visual Acuity in the Study Eye (or Eyes) at Week 36 Compared to Baseline
Description: as for outcome 2
Time Frame: Baseline and Week 36
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: eyes
Arm/Group | Gevokizumab
Number analyzed (Participants) | 6
Number analyzed (eyes) | 6
ETDRS letters | 1.83 (5.12)

12. Secondary Outcome: Mean Change in Visual Acuity in the Study Eye (or Eyes) at Week 40 Compared to Baseline
Description: as for outcome 2
Time Frame: Baseline and Week 40
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: eyes
Arm/Group | Gevokizumab
Number analyzed (Participants) | 6
Number analyzed (eyes) | 6
ETDRS letters | 2.67 (5.39)

13. Secondary Outcome: Mean Change in Visual Acuity in the Study Eye (or Eyes) at Week 52 Compared to Baseline
Description: as for outcome 2
Time Frame: Baseline and Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: eyes
Arm/Group | Gevokizumab
Number analyzed (Participants) | 6
Number analyzed (eyes) | 6
ETDRS letters | 0.17 (6.43)

14. Secondary Outcome: Mean Change in Visual Acuity in the Study Eye (or Eyes) at Week 52A Compared to Baseline
Description: This visit represents the beginning of the as-needed 2nd Extension Phase at Week 52. If eligible, participants continued with injections at Wks 52, 54, 58 and 62.
  Visual acuity was measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol. Acuity is measured as letters read on an ETDRS eye chart and the letters read equate to Snellen measurements. For example, if a participant reads between 84 and 88 letters, the equivalent Snellen measurement is 20/20.
Time Frame: Baseline and Week 52A
Population: Eight participants were active from Baseline to Week 28. Of the 8 active participants, one participant had two study eyes and was active to Week 28. Two participants did not continue past Week 28 due to insufficient therapeutic response. Six participants were active from Week 32 to Week 52. Three participants were active from Week 52 to study end.
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: eyes
Arm/Group | Gevokizumab
Number analyzed (Participants) | 3
Number analyzed (eyes) | 3
ETDRS letters | -8.00 (13.45)

15. Secondary Outcome: Mean Change in Visual Acuity in the Study Eye (or Eyes) at Week 54 Compared to Baseline
Description: as for outcome 2
Time Frame: Baseline and Week 54
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: eyes
Arm/Group | Gevokizumab
Number analyzed (Participants) | 3
Number analyzed (eyes) | 3
ETDRS letters | -0.67 (6.03)

16. Secondary Outcome: Mean Change in Visual Acuity in the Study Eye (or Eyes) at Week 58 Compared to Baseline
Description: as for outcome 2
Time Frame: Baseline and Week 58
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: eyes
Arm/Group | Gevokizumab
Number analyzed (Participants) | 3
Number analyzed (eyes) | 3
ETDRS letters | -1.33 (6.51)

17. Secondary Outcome: Mean Change in Visual Acuity in the Study Eye (or Eyes) at Week 62 Compared to Baseline
Description: as for outcome 2
Time Frame: Baseline and Week 62
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: eyes
Arm/Group | Gevokizumab
Number analyzed (Participants) | 3
Number analyzed (eyes) | 3
ETDRS letters | -1.33 (5.03)

18. Secondary Outcome: Mean Change in Visual Acuity in the Study Eye (or Eyes) at Final Safety Visit Compared to Baseline
Description: as for outcome 2
Time Frame: Baseline and Final Visit
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: eyes
Arm/Group | Gevokizumab
Number analyzed (Participants) | 3
Number analyzed (eyes) | 3
ETDRS letters | -2.00 (4.36)

19. Secondary Outcome: Mean Change in Intraocular Pressure in the Study Eye (or Eyes) at Week 2 Compared to Baseline
Description: Intraocular pressure (IOP) is measured in millimeters of mercury (mmHg).
Time Frame: Baseline and Week 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | Gevokizumab
Number analyzed (Participants) | 8
Number analyzed (eyes) | 9
mmHg | 0.67 (1.94)

20. Secondary Outcome: Mean Change in Intraocular Pressure in the Study Eye (or Eyes) at Week 4 Compared to Baseline
Description: Intraocular pressure (IOP) is measured in millimeters of mercury (mmHg).
Time Frame: Baseline and Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | Gevokizumab
Number analyzed (Participants) | 8
Number analyzed (eyes) | 9
mmHg | 0.67 (3.04)

21. Secondary Outcome: Mean Change in Intraocular Pressure in the Study Eye (or Eyes) at Week 8 Compared to Baseline
Description: Intraocular pressure (IOP) is measured in millimeters of mercury (mmHg).
Time Frame: Baseline and Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | Gevokizumab
Number analyzed (Participants) | 8
Number analyzed (eyes) | 9
mmHg | 1.11 (1.69)

22. Secondary Outcome: Mean Change in Intraocular Pressure in the Study Eye (or Eyes) at Week 12 Compared to Baseline
Description: Intraocular pressure (IOP) is measured in millimeters of mercury (mmHg).
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | Gevokizumab
Number analyzed (Participants) | 8
Number analyzed (eyes) | 9
mmHg | 1.00 (3.67)

23. Secondary Outcome: Mean Change in Intraocular Pressure in the Study Eye (or Eyes) at Week 16 Compared to Baseline
Description: Intraocular pressure (IOP) is measured in millimeters of mercury (mmHg).
Time Frame: Baseline and Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | Gevokizumab
Number analyzed (Participants) | 8
Number analyzed (eyes) | 9
mmHg | 1.56 (2.07)

24. Secondary Outcome: Mean Change in Intraocular Pressure in the Study Eye (or Eyes) at Week 20 Compared to Baseline
Description: Intraocular pressure (IOP) is measured in millimeters of mercury (mmHg).
Time Frame: Baseline and Week 20
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | Gevokizumab
Number analyzed (Participants) | 8
Number analyzed (eyes) | 9
mmHg | 1.33 (2.00)

25. Secondary Outcome: Mean Change in Intraocular Pressure in the Study Eye (or Eyes) at Week 24 Compared to Baseline
Description: Mean Change in Intraocular pressure (IOP) is measured and reported as change in IOP between baseline and 24 weeks in millimeters of mercury (mmHg).
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | Gevokizumab
Number analyzed (Participants) | 8
Number analyzed (eyes) | 9
mmHg | 0.78 (2.33)

26. Secondary Outcome: Mean Change in Intraocular Pressure in the Study Eye (or Eyes) at Week 28 Compared to Baseline
Description: Intraocular pressure (IOP) is measured in millimeters of mercury (mmHg).
Time Frame: Baseline and Week 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | Gevokizumab
Number analyzed (Participants) | 8
Number analyzed (eyes) | 9
mmHg | 1.11 (2.26)

27. Secondary Outcome: Mean Change in Intraocular Pressure in the Study Eye (or Eyes) at Week 32 Compared to Baseline
Description: Intraocular pressure (IOP) is measured in millimeters of mercury (mmHg).
Time Frame: Baseline and Week 32
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | Gevokizumab
Number analyzed (Participants) | 6
Number analyzed (eyes) | 6
mmHg | 2.67 (1.75)

28. Secondary Outcome: Mean Change in Intraocular Pressure in the Study Eye (or Eyes) at Week 36 Compared to Baseline
Description: Intraocular pressure (IOP) is measured in millimeters of mercury (mmHg).
Time Frame: Baseline and Week 36
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | Gevokizumab
Number analyzed (Participants) | 6
Number analyzed (eyes) | 6
mmHg | 2.17 (1.72)

29. Secondary Outcome: Mean Change in Intraocular Pressure in the Study Eye (or Eyes) at Week 40 Compared to Baseline
Description: Intraocular pressure (IOP) is measured in millimeters of mercury (mmHg).
Time Frame: Baseline and Week 40
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | Gevokizumab
Number analyzed (Participants) | 6
Number analyzed (eyes) | 6
mmHg | 0.50 (1.52)

30. Secondary Outcome: Mean Change in Intraocular Pressure in the Study Eye (or Eyes) at Week 52 Compared to Baseline
Description: Intraocular pressure (IOP) is measured in millimeters of mercury (mmHg).
Time Frame: Baseline and Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | Gevokizumab
Number analyzed (Participants) | 6
Number analyzed (eyes) | 6
mmHg | 1.83 (2.79)

31. Secondary Outcome: Mean Change in Intraocular Pressure in the Study Eye (or Eyes) at Week 52A Compared to Baseline
Description: This visit represents the beginning of the as-needed 2nd Extension Phase at Week 52. If eligible, participants continued with injections at Wks 52, 54, 58 and 62.
  Intraocular pressure (IOP) is measured in millimeters of mercury (mmHg).
Time Frame: Baseline and Week 52A
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | Gevokizumab
Number analyzed (Participants) | 3
Number analyzed (eyes) | 3
mmHg | -0.67 (2.08)

32. Secondary Outcome: Mean Change in Intraocular Pressure in the Study Eye (or Eyes) at Week 54 Compared to Baseline
Description: Intraocular pressure (IOP) is measured in millimeters of mercury (mmHg).
Time Frame: Baseline and Week 54
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | Gevokizumab
Number analyzed (Participants) | 3
Number analyzed (eyes) | 3
mmHg | 1.33 (4.16)

33. Secondary Outcome: Mean Change in Intraocular Pressure in the Study Eye (or Eyes) at Week 58 Compared to Baseline
Description: Intraocular pressure (IOP) is measured in millimeters of mercury (mmHg).
Time Frame: Baseline and Week 58
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | Gevokizumab
Number analyzed (Participants) | 3
Number analyzed (eyes) | 3
mmHg | 1.33 (3.21)

34. Secondary Outcome: Mean Change in Intraocular Pressure in the Study Eye (or Eyes) at Week 62 Compared to Baseline
Description: Intraocular pressure (IOP) is measured in millimeters of mercury (mmHg).
Time Frame: Baseline and Week 62
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | Gevokizumab
Number analyzed (Participants) | 3
Number analyzed (eyes) | 3
mmHg | 0.67 (1.53)

35. Secondary Outcome: Mean Change in Intraocular Pressure in the Study Eye (or Eyes) at Final Safety Visit Compared to Baseline
Description: Intraocular pressure (IOP) is measured in millimeters of mercury (mmHg).
Time Frame: Baseline and Final Visit
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | Gevokizumab
Number analyzed (Participants) | 3
Number analyzed (eyes) | 3
mmHg | 1.33 (2.08)

36. Secondary Outcome: Number of Participants With Loss of ≥ 15 Early Treatment Diabetic Retinopathy Study (ETDRS) Letters
Description: as for outcome 2
Time Frame: Post-injection through study completion, up to 78 weeks per participant
Population: as for outcome 14
Measure: Number; unit: participants
Units Other Than Participants: eyes
Arm/Group | Gevokizumab
Number analyzed (Participants) | 8
Number analyzed (eyes) | 9
participants | 0

37. Secondary Outcome: Changes in Scleral Grading From Baseline to Week 52
Description: Scleral inflammation was summarized on an ordinal scale as either none, minimal/trace, mild, moderate, severe or necrotizing inflammation in the four quadrants of the study eye (superonasal [SN], superotemporal [ST], inferotemporal [IT], and inferonasal [IN]) for each participant at each visit. The exact change from Baseline to Week 52 for each participant (such as from mild to severe) cannot be quantified; therefore, we chose not to report due to the difficulty of reporting a quantitative change in each quadrant for each participant within the limited parameters allowed by PRS.
Time Frame: Baseline and Week 52
Population: The exact change from Baseline to Week 52 for each participant (such as from mild to severe) cannot be quantified; therefore, we chose not to report due to the difficulty of reporting a quantitative change in each quadrant for each participant within the limited parameters allowed by PRS.
Arm/Group | Gevokizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline until study completion, up to 78 weeks (wks) per participant. Participants in the 2nd extension phase had a final safety visit at least 16 wks following their last injection in the 2nd extension phase at Wk 62.
Arm/Group | Gevokizumab
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gevokizumab (N=8)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Bacterial test (Investigations) | 1 (1)
Biopsy skin (Investigations) | 1 (1)
Corneal thinning (Eye disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Foreign body in eye (Injury, poisoning and procedural complications) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Hemoglobin urine present (Investigations) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (3)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Ocular hyperaemia (Eye disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritis generalized (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (2)
Renal failure (Renal and urinary disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Scleral thinning (Eye disorders) | 1 (2)
Sinusitis (Infections and infestations) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (2)
Injection site discomfort (General disorders) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No